CLINICAL TRIAL: NCT00004231
Title: Phase II Study of Multimodality Therapy in Mantle Cell Lymphoma
Brief Title: Combination Chemotherapy, Bone Marrow or Peripheral Stem Cell Transplantation, and/or Biological Therapy in Treating Patients With Stage III or Stage IV Mantle Cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: NU 96H3; NU-96H3; NCI-G99-1659
Record Dates: First submitted 2000-01-28; First posted 2003-01-27 (Estimated); Last update posted 2012-06-06 (Estimated); Status verified 2012-05

CONDITIONS: Lymphoma
Keywords: stage III mantle cell lymphoma; stage IV mantle cell lymphoma; recurrent mantle cell lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Mantle-Cell | interventions — aldesleukin; Filgrastim; Interferon-alpha; Busulfan; Cyclophosphamide; Cytarabine; Doxorubicin; Leucovorin; Methotrexate; Prednisone; Teniposide; Vincristine; Peripheral Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: aldesleukin
Biological: filgrastim
Biological: recombinant interferon alfa
Drug: busulfan
Drug: cyclophosphamide
Drug: cytarabine
Drug: doxorubicin hydrochloride
Drug: leucovorin calcium
Drug: methotrexate
Drug: prednisone
Drug: teniposide
Drug: vincristine sulfate
Procedure: allogeneic bone marrow transplantation
Procedure: autologous bone marrow transplantation
Procedure: peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining chemotherapy with peripheral stem cell or bone marrow transplantation may allow the doctor to give higher doses of chemotherapy drugs and kill more cancer cells. Biological therapies use different ways to stimulate the immune system and stop cancer cells from growing.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy followed by bone marrow or peripheral stem cell transplantation and/or biological therapy in treating patients who have stage III, stage IV, or recurrent mantle cell lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the toxicities of combination chemotherapy followed by allogeneic or autologous bone marrow transplantation or peripheral blood stem cell transplantation and/or interferon and interleukin therapy in patients with refractory or stage III or IV mantle cell lymphoma.
* Determine the complete response rate in these patients after these treatments.
* Evaluate the prognostic factors in this patient population.

OUTLINE: This is a multicenter study.

Patients receive induction chemotherapy consisting of cyclophosphamide IV, doxorubicin IV, and teniposide IV over 2 hours on day 1, oral prednisone on days 1-5, vincristine IV and methotrexate IV over 2 hours on day 21, cytarabine IV over 2 hours every 12 hours for a total of 2 doses on day 22, and oral leucovorin calcium every 6 hours beginning on day 22 and continuing until methotrexate levels recover. Treatment repeats every 42 days for 2 courses. Patients achieving complete response or partial response receive an additional course of induction therapy. Patients achieving maximal response following 2 courses of induction chemotherapy undergo transplantation.

Patients under 50 years with an HLA matched donor undergo allogeneic bone marrow transplantation (BMT). Patients receive busulfan IV every 6 hours for a total of 14 doses beginning on day -8 and continuing for 3.5 days. At 24 hours following the last dose of busulfan, patients receive cyclophosphamide IV over 2 hours daily for 2 days. Patients receive allogeneic bone marrow infusion on day 0.

Patients under 50 years with no HLA matched donor or patients 50-65 years old undergo autologous bone marrow or peripheral blood stem cell (PBSC) transplantation. Patients undergo PBSC mobilization following completion of cyclophosphamide, doxorubicin, and teniposide portion of induction therapy of course 3. Patients receive cytokines subcutaneously (SQ) beginning 2 days following chemotherapy and continuing through PBSC collection. If insufficient stem cells are collected and there is negative bone marrow involvement, patients undergo bone marrow harvest. Patients receive a conditioning regimen consisting of busulfan and cyclophosphamide as for allogeneic BMT. Patients receive autologous bone marrow or PBSC infusion on day 0 and filgrastim (G-CSF) SQ beginning on day 0 and continuing until blood counts recover. Following blood count recovery, patients receive maintenance therapy consisting of interferon alfa SQ and interleukin-2 SQ daily over 5 consecutive days for 4 weeks. Treatment repeats every 8 weeks for 2 courses.

Patients 65 years or older achieving complete or partial response to induction chemotherapy receive maintenance therapy as for autologous BMT. Patients achieving partial response may receive an additional 4th course of induction therapy prior to maintenance therapy.

Patients are followed at 30 days post transplant, every 3 months for 1 year, and then at least every 6 months for 2 years.

PROJECTED ACCRUAL: A total of 15-48 patients will be accrued for this study over 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed stage III, IV, or recurrent mantle cell lymphoma

  * CD5 positive OR
  * Evidence of bcl-1 oncogene overexpression
* Measurable or evaluable disease with at least one of the following:

  * Clear cut radiographic findings
  * Clearly defined bidimensional defect or mass at least 2 cm in diameter on radionuclide or CT scan
  * Enlarged spleen extending at least 2 cm below costal margin with lymphomatous involvement only
  * Enlarged liver with proof of lymphoma by biopsy
* CNS involvement allowed
* Fully HLA matched donor for allogeneic transplantation

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-3

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Bilirubin no greater than 3.0 mg/dL

Renal:

* Creatinine no greater than 2.0 mg/dL

Cardiovascular:

* No significant cardiac disease

Other:

* No other prior malignancies except previously treated nonmelanoma skin cancer or carcinoma in situ of the cervix
* No other medical problems that would preclude study
* HIV negative
* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* See Disease Characteristics

Chemotherapy:

* See Disease Characteristics
* Prior chemotherapy, including doxorubicin, allowed

Endocrine therapy:

* See Disease Characteristics
* Prior steroids allowed

Radiotherapy:

* See Disease Characteristics
* Prior radiotherapy allowed excluding the indicator lesions

Surgery:

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-10; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leo I. Gordon, MD, Study Chair — Robert H. Lurie Cancer Center
Locations (1):
- Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois, United States

REFERENCES:
- [Result] Evens AM, Winter JN, Hou N, Nelson BP, Rademaker A, Patton D, Singhal S, Frankfurt O, Tallman MS, Rosen ST, Mehta J, Gordon LI. A phase II clinical trial of intensive chemotherapy followed by consolidative stem cell transplant: long-term follow-up in newly diagnosed mantle cell lymphoma. Br J Haematol. 2008 Feb;140(4):385-93. doi: 10.1111/j.1365-2141.2007.06908.x. Epub 2007 Dec 19. PMID 18162124